CLINICAL TRIAL: NCT05787314
Title: Low Glycemic Index Diet Effects in Obesity With Insulin Resistance
Brief Title: Effect of Low Glycemic Index Diet on Biochemical Parameters and Body Image in Obesity With Insulin Resistance: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Mesut Karahan, Assoc. Prof., Uskudar University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UskudarUBesYA02
Record Dates: First submitted 2023-03-12; First posted 2023-03-28 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Low Glycemic Load Diet; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Different nutrition programs were applied to obese individuals divided into control and experimental groups. While the experimental group was given a healthy/balanced nutrition program containing carbohydrates and aimed to lose weight, a nutritional program that was balanced and aimed to lose weight but did not make any classification was applied to the control group. At the end of 8 weeks, biochemical parameters and scales were compared.
Masking Description: prospective, two-arm randomized-controlled trial, Researchers who have no knowledge about group allocation and study's objectives, will collected the post-intervention data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Diet (Experimental): 1. For the Control Diet, a medical nutrition therapy with calorie and fat content was prepared to ensure weight loss of individuals without considering the glycemic index.
  2. The aim of this diet is to achieve weight loss, but not to focus on the content of carbohydrates. 3) In the macro element distribution of the CD, 50-55% carbohydrates, 10-15% protein and 20-25% fat distribution Other name (CD Group)
  Interventions: Behavioral: Low Glycemic Index Diet

INTERVENTIONS:
Behavioral: Low Glycemic Index Diet — 1. Participants who came to the hospital for control and were interested in the study contacted the study researchers and eligibility was determined through face-to-face interviews. Potential participants were invited to a screening visit to verify eligibility.
  2. The LGID program was initiated as an outpatient treatment in patients who applied to a dietitian. 3) Medium and high GI carbohydrates (GI > 55) were excluded from the diet and only low GI (GI < 50) foodstuffs were allowed. 4) A list of low glycemic index foods were given to the patients. In addition, a list of foods to avoid (medium and high glycemic index) is provided.
  Other Names: LGID Group

SUMMARY:
To examine how a low glycemic index diet (LGID) changes biochemical parameters, body measurements, and body image perception in obese individuals with insulin resistance. Obesity groups with insulin resistance who received a control diet (CD) and a LGID will be compared with each other in terms of biochemical parameters, body image perception and body measurements. In addition, each group will be compared with the start and end measurements over the same values.

DETAILED DESCRIPTION:
The main purpose of this study is to determine the effect of LGID on body image perception, biochemical parameters and body measurements in obese individuals with insulin resistance.

Sub-objectives of the study;

Determination of the effect of LGID on fasting blood glucose, fasting insulin level and HOMA-IR levels compared to CD.

Determination of the effect of LGID on body weight, fat mass, muscle mass, body muscle ratio and body mass index (BMI) compared to CD.

Determination of the effect of LGID on body image perception status compared to CD.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 24 kg/m2, or the either one (fat mass ≧ 30% or waistline > 80 cm)
* Can provide informed consent
* Can be contacted by telephone
* Waist circumference > 90 cm for men and > 80 cm for women

Exclusion Criteria:

* Pregnancy or lactation
* Active or suspected chronic infection
* Treatment affecting insulin sensitivity
* A secondary disease state (Cardiovascular disease, cancer, psychiatric, etc.)
* Any weight loss operation (gastric bypass, gastric balloon, etc.)
* A special nutritional program (cancer, kidney disease, etc.)
* Using any food supplement or medication known to affect whole body metabolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Homeostatic Model Assessment for Insulin Resistance | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) index was obtained by the following formula: fasting glucose (mg/dl/18) x fasting insulin (U/mL)/22.5.
  A HOMA-IR index >2.5 is in favor of Insulin Resistance (IR).
Cholesterol | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Blood samples were collected after an overnight fast by using 10 mL plain tubes. Lipid profile was measured by using Cholesterol Kits and total cholesterol levels were measured using the sum of the LDL and HDL plus one-fifth of triglyceride levels.
Fasting plasma glucose | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Fasting plasma glucose (FPG) levels were determined by taking a blood sample from participants who have fasted for at least 8 hours, Fasting glucose is between 75-95 mg/dL (4.2-5.3 mmol/L).
Fasting insulin level | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Fasting insulin is between 18-48 pmol/L.
Body weight | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Body weight was measured in kilograms.
Body muscle ratio | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Body muscle ratio as assessed by bioelectrical impedance analysis -- whole body composition was evaluated.
Body muscle mass, kg | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Body muscle mass as assessed by bioelectrical impedance analysis -- whole body composition was evaluated.
Body mass index | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Body mass index (BMI)=weight/(height)^2
Body fat mass, kg | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Body fat mass as assessed by bioelectrical impedance analysis -- whole body composition was evaluated.
Body fat ratio | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  Body fat ratio as assessed by bioelectrical impedance analysis -- whole body composition was evaluated.

SECONDARY OUTCOMES:
Assessment of body image scale | Changes within and between groups are evaluated on the start and last day of the intervention (day 120).
  The body image scale (BIS) includes 10 items, and was developed to briefly and comprehensively assess the affective (e.g., feeling self-conscious), behavioral (e.g., difficulty in looking at the naked body), and cognitive (e.g., satisfaction with appearance) aspects of body image in patients. It is a 4-point scale (0 = not at all and 3 = very much), and the final score is the sum of scores for 10 items, ranging from 0 to 30, with a lower score representing a better body image.

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar University, Istanbul, Turkey (Türkiye)